CLINICAL TRIAL: NCT01598311
Title: A Randomized, Double-Blinded, Active-Controlled Study of CB-183,315 in Patients With Clostridium Difficile Associated Diarrhea
Brief Title: A Study of CB-183,315 in Participants With Clostridium Difficile Associated Diarrhea (MK-4261-006)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4261-006; LCD-CDAD-11-06 (Other: Cubist Protocol Number); MK-4261-006 (Other: Merck Protocol Number); 2012-000252-34 (EudraCT Number)
Record Dates: First submitted 2012-05-10; First posted 2012-05-15 (Estimated); Results first posted 2018-02-27 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Clostridium Difficile Infection
Keywords: CDAD; Clostridium difficile Associated Diarrhea; CDI; Clostridium difficile Infection; Diarrhea
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — CB-183,315; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CB-183,315 (Experimental): Participants took CB-183,315 250 mg twice daily (b.i.d.) and placebo capsules b.i.d. by mouth for 10 days.
  Interventions: Drug: CB-183,315; Drug: Placebo
- Vancomycin (Active Comparator): Participants took vancomycin 125 mg four times daily (q.i.d.) by mouth for 10 days.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: CB-183,315 — CB-183,315 250 mg white coated tablet over-encapsulated in a size 00 opaque hard gelatin capsule.
  Other Names: Surotomycin
  Arms: CB-183,315
Drug: Vancomycin — Vancomycin hydrochloride 125 mg capsule over-encapsulated in size 00 opaque hard gelatin capsule.
  Arms: Vancomycin
Drug: Placebo — Placebo size 00 opaque hard gelatin capsules.
  Arms: CB-183,315

SUMMARY:
A total of 608 participants with Clostridium Difficile Associated Diarrhea (CDAD) will participate in this study; participants will receive either oral vancomycin or CB-183,315 in a blinded fashion. Treatment will last for 10 days and participants will be followed up for at least 40 days and a maximum of 100 days. The purpose of this study is to evaluate how well CB-183,315 treats CDAD as compared to vancomycin.

ELIGIBILITY:
Inclusion Criteria:

* Is able to read and sign a consent form;
* Is from ≥18 to <90 years of age;
* Has diarrhea, at least 3 times during one day, or 200 mL or liquid stool if using a rectal device;
* Tests positive for Clostridium difficile;
* If female, must not be pregnant or nursing and take appropriate measures to not get pregnant during the study.

Exclusion Criteria:

* Has toxic megacolon and/or known small bowel ileus;
* Has received treatment with intravenous immune globulin (IVIG) within the past 30 days;
* Has received treatment with a fecal transplant within 7 days, and/or if the doctor anticipates to give the participant a fecal transplant during the study;
* Has received a certain amount of antibacterial therapy specific for current CDAD, unless it is not working;
* Has received an investigational vaccine against Clostridium difficile;
* Has received an investigational product containing monoclonal antibodies against toxin A or B within 180 days;
* Has more than 2 episodes of CDAD within 90 days;
* Has had major gastrointestinal (GI) surgery (i.e. significant bowel resection) within 3 months (this does not include appendectomy or cholecystectomy);
* Has a history of prior inflammatory bowel disease: ulcerative colitis, Crohn's disease, or microscopic colitis;
* Is unable to discontinue loperamide, diphenoxylate/atropine, or cholestyramine during the duration of the study;
* Is unable to discontinue opiate treatment unless on a stable dose;
* Has known positive stool cultures for other enteropathogens including but not limited to Salmonella, Shigella, and Campylobacter;
* Has had stool studies positive for pathogenic ova and/or parasites;
* Has an intolerance or hypersensitivity to daptomycin and/or vancomycin;
* Has a life-threatening illness at the time of enrollment;
* Has poor concurrent medical risks that in the opinion of the Investigator the participant should not enroll;
* Has received an investigational drug or participated in any experimental procedure within 1 month;
* Has human immunodeficiency virus (HIV), a cluster of differentiation (CD) 4 count <200 cells/mm^3 within 6 months of start of study therapy;
* Anticipates that certain antibacterial therapy for a non-CDAD infection will be required for >7 days;
* Is unable to discontinue Saccharomyces or similar probiotic;
* Is on a concurrent intensive induction chemotherapy, radiotherapy, or biologic treatment for active malignancy;
* Is unable to comply with the protocol requirements;
* Has any condition that, in the opinion of the Investigator, might interfere;
* Is not expected to live for less than 8 weeks.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2012-05-16 (Actual); Primary Completion 2015-07-26 (Actual); Study Completion 2015-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Daley P, Louie T, Lutz JE, Khanna S, Stoutenburgh U, Jin M, Adedoyin A, Chesnel L, Guris D, Larson KB, Murata Y. Surotomycin versus vancomycin in adults with Clostridium difficile infection: primary clinical outcomes from the second pivotal, randomized, double-blind, Phase 3 trial. J Antimicrob Chemother. 2017 Dec 1;72(12):3462-3470. doi: 10.1093/jac/dkx299. PMID 28961905
- [Derived] Cheknis A, Devaris D, Chesnel L, Dale SE, Nary J, Sambol SP, Citron DM, Goering RV, Johnson S. Characterization of Clostridioides difficile isolates recovered from two Phase 3 surotomycin treatment trials by restriction endonuclease analysis, PCR ribotyping and antimicrobial susceptibilities. J Antimicrob Chemother. 2020 Nov 1;75(11):3120-3125. doi: 10.1093/jac/dkaa297. PMID 32747931

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled adult participants with Clostridium Difficile associated diarrhea (CDAD) at 104 study centers in North America, Asia-Pacific, and South America.
Groups:
- CB-183,315: Participants took CB-183,315 250 mg twice daily (b.i.d.) and placebo b.i.d. by mouth for 10 days.
Period: Overall Study
Arm/Group | CB-183,315 | Vancomycin
Started (Randomized) | 303 | 305
Treated (Safety Population) | 294 | 301
Treated and Confirmed CDAD (mMITT Population) | 285 | 292
Completed | 256 | 244
Not Completed | 47 | 61
Not completed — Physician Decision | 4 | 5
Not completed — Adverse Event | 9 | 13
Not completed — Lost to Follow-up | 7 | 12
Not completed — Withdrawal by Subject | 9 | 13
Not completed — No reason provided. | 0 | 5
Not completed — Randomized but never treated | 8 | 5
Not completed — Treated but no confirmed CDAD | 9 | 8
Not completed — Assigned to CB but received vancomycin | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all randomized and treated participants with a confirmed CDAD diagnosis (microbiological modified intent-to-treat [mMITT] population).
Groups:
- CB-183,315: Participants took CB-183,315 250 mg b.i.d. and placebo b.i.d. by mouth for 10 days.
- Vancomycin: Participants took vancomycin 125 mg q.i.d. by mouth for 10 days.
- Total: Total of all reporting groups
Arm/Group | CB-183,315 | Vancomycin | Total
Number analyzed (Participants) | 285 | 292 | 577
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (18.3) | 56.5 (18.3) | 57.1 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 194 | 367
  Male | 112 | 98 | 210

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Percentage of Participants Meeting Clinical Response Criteria for Cure at End of Treatment (EOT)
Description: The percentage of participants considered "cured" (i.e., ≤2 loose stools per 24 hour period for at least 2 consecutive days and no need for additional antibiotics during the 3 days following EOT) was determined in the mMITT population. A CDAD diagnosis was defined as: 1) diarrhea with a minimum of 3 unformed bowel movements (UBM) or >200 mL volume of stool for participants with a collection device (e.g., rectal tube or colostomy bag) over 24 hours; and 2) a positive result for Clostridium difficile toxin by enzyme immunoassay (EIA), polymerase chain reaction (PCR), or a cell culture cytotoxin neutralization assay. Percentages were first stratified according to age (<75 or ≥75 years) and number of previous CDAD episodes (0 or ≥1) and constructed using Mehrotra-Railkar continuity-corrected minimum-risk stratum weights, and the weighted averages were then derived across strata in order to calculate the adjusted percentage.
Time Frame: Up to 3 days after EOT (up to Day 13)
Population: The analysis population consists of all randomized and treated participants with a confirmed CDAD diagnosis (mMITT population).
Measure: Number (95% Confidence Interval); unit: Adjusted percentage of participants
Arm/Group | CB-183,315 | Vancomycin
Number analyzed (Participants) | 285 | 292
Adjusted percentage of participants | 83.4 [78.7 to 87.2] | 82.1 [77.2 to 85.9]
Statistical Analysis 1: Comparison: CB-183,315 vs Vancomycin; Test type: Non-Inferiority — Non-inferiority was declared when the lower bound of the 95% CI for the difference in adjusted percentage of cured subjects was > -10%; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-4.9 to 7.6]

2. Secondary Outcome: Number of Clinical Failure Events up to Day 40
Description: The total number of clinical failure events, which included treatment failure, CDAD recurrence, death, or being lost to follow-up, occurring during each time period was determined in each arm.
Time Frame: Up to 30 days after EOT (up to Day 40)
Population: as for outcome 1
Measure: Number; unit: Number of Failure Events
Arm/Group | CB-183,315 | Vancomycin
Number analyzed (Participants) | 285 | 292
Number of Failure Events
  Day 0 to Day 13 | 48 | 54
  Day 14 to Day 24: number analyzed (Participants) | 237 | 238
  Day 14 to Day 24 | 42 | 49
  Day 25 to Day 35: number analyzed (Participants) | 195 | 189
  Day 25 to Day 35 | 11 | 11
  Day 36 to Day 40: number analyzed (Participants) | 184 | 178
  Day 36 to Day 40 | 2 | 2

3. Secondary Outcome: Adjusted Percentage of Participants With Sustained Clinical Response at End of Study
Description: The percentage of participants with sustained clinical response was determined for each arm. Sustained clinical response was declared when participants had a clinical outcome of cure at EOT, did not experience any CDAD recurrence, did not die, were not lost to follow-up, and did not have the end of study visit prior to Day 40. Percentages were first stratified according to age (<75 or ≥75 years) and number of previous CDAD episodes (0 or ≥1) and constructed using Mehrotra-Railkar continuity-corrected minimum-risk stratum weights, and the weighted averages were then derived across strata in order to calculate the adjusted percentage.
Time Frame: Up to 40 days after EOT (up to Day 50)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Adjusted percentage of participants
Arm/Group | CB-183,315 | Vancomycin
Number analyzed (Participants) | 285 | 292
Adjusted percentage of participants | 63.3 [57.7 to 68.7] | 59.0 [53.4 to 64.5]
Statistical Analysis 1: Comparison: CB-183,315 vs Vancomycin; Test type: Superiority — Superiority was declared if the lower bound of the 95% CI of the adjusted difference in sustained response was > 0; Mean Difference (Final Values) = 4.3, 95% CI 2-sided [-3.6 to 12.2]

4. Primary Outcome: Percentage of Participants Experiencing an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 30 days after EOT (up to Day 40)
Population: The analysis population consists of all randomized and treated participants (Safety Population).
Measure: Number; unit: Percentage of Participants
Arm/Group | CB-183,315 | Vancomycin
Number analyzed (Participants) | 294 | 301
Percentage of Participants | 52.4 | 60.1

5. Primary Outcome: Percentage of Participants Discontinuing From Study Treatment Due to an AE
Description: as for outcome 4
Time Frame: Up to EOT (up to Day 10)
Population: The analysis population consists of all randomized and treated participants (Safety Population).
Measure: Number; unit: Percentage of Participants
Arm/Group | CB-183,315 | Vancomycin
Number analyzed (Participants) | 294 | 301
Percentage of Participants | 3.7 | 3.0

ADVERSE EVENTS:
Time Frame: All AEs were collected up to Day 13; only serious AEs (SAEs) and drug-related AEs were collected up to Day 50.
Description: The analysis population consists of all randomized participants who received ≥1 dose of study drug.
Arm/Group | CB-183,315 | Vancomycin
All-Cause Mortality (participants affected / at risk) | 9/294 | 11/301
Serious Adverse Events (participants affected / at risk) | 33/294 | 39/301
Other Adverse Events (participants affected / at risk) | 53/294 | 72/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CB-183,315 (N=294) | Vancomycin (N=301)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 4 (4) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Heart transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 2 (2)
Serratia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CB-183,315 (N=294) | Vancomycin (N=301)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 22 (23)
Nausea (Gastrointestinal disorders) | 25 (25) | 23 (23)
Headache (Nervous system disorders) | 31 (33) | 36 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No